CLINICAL TRIAL: NCT00604422
Title: Evaluation of the PillCam™ Colon Capsule Endoscopy (PCCE) in Detection & Classification of Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-107
Record Dates: First submitted 2008-01-24; First posted 2008-01-30 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2010-03

CONDITIONS: Colonic Disease; Ulcerative Colitis
Keywords: Colonic disease; Ulcerative colitis; suspected or known colonic disease
MeSH Terms: conditions — Colonic Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Subjects that are indicated for standard colonoscopy due to suspected or known Ulcerative colitis disease

SUMMARY:
To evaluate the ability of the PillCam® Colon Capsule Endoscope to detect and classify Ulcerative colitis

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a disorder of unknown origin that may be characterized by acute and chronic inflammation of the colon. The extent of the colonic mucosal inflammation varies among individuals, but the disease almost always involves the rectum. Ulcerative colitis has required evaluation by colonoscopy to determine the extent and severity of the disease. The PillCam platform offers an alternative approach for endoscopic visualization of the colon using capsule endoscopy, a swallowable device which contains imagers, light sources, a power source and a RF transmitter. Advantages of the PillCam platform include the elimination of the need for conscious sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure . Furthermore, compared to standard colonoscopy, the PillCam platform may be more readily accepted by the subjects, thereby improving subjects' willingness to undergo a diagnostic evaluation of the colon.

The PillCam® SB capsule (formerly M2A® Capsule) that was FDA-approved in August 2001 for small bowel evaluation has been ingested to date by more than 700,000 people worldwide and is well accepted by patients and physicians as well as the professional societies. However, adequate visualization of the colon cannot be achieved with the standard PillCam™ SB capsule because of the anatomical and physiological properties of the colon which are significantly different than the small bowel. Moreover, other issues that limit the evaluation of the colonic mucosa by the standard PillCam™ SB procedure include an unsatisfactory level of colon cleanliness and slow progression of the PillCam™ SB capsule through the colon during the desired examination time. Therefore, the development and introduction of a specially designed, customized colon capsule combined with a dedicated capsule colonoscopy procedure protocol will allow for more efficient evaluation of the colonic mucosa. Further details of the PillCam® Colon Capsule Endoscope (PCCE) can be found in the device description section.

In previous studies, the PillCam colon platform has been shown to be safe and to be able to demonstrate colon polyps and cancers. This study is an extension to a trial evaluating the use of PCCE in ulcerative colitis that has already been completed in Hong Kong (n=40). This study is designed to assess the ability of the capsule to accurately detect inflammatory lesions and thus classifying the extent and severity of disease in subjects with ulcerative colitis in comparison to traditional colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-70
* Suspected or known ulcerative colitis patients

Exclusion Criteria:

* Subject has dysphagia
* Subject has congestive heart failure
* Subject who can not tolerate bowel preparation
* Poor bowel preparation
* Subject has renal insufficiency
* Subject is known or is suspected to suffer from intestinal obstruction.
* Subject has a cardiac pacemaker or other implanted electro-medical devices.
* Subject is pregnant
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Subject suffers from life threatening conditions
* Subject is currently participating in another clinical study
* Subject has constipation (less than 3 bowel movements/week)
* Subject has known slow gastric emptying time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that are indicated for standard colonoscopy due to suspected or known Ulcerative colitis disease
  The study population will consist of subjects who fulfill all the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2007-04; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Agreement level between capsule and colonoscopy in classifying colitis into the above (see section 3.1) categories. | within 7 days

SECONDARY OUTCOMES:
Number, type and severity of adverse events with both PCCE and standard colonoscopy | Within 7 days
Accuracy parameters for detecting active UC | within 7 days
Disease severity scoring index for both PCCE and .standard colonoscopy | within 7 days
Colon cleansing level score for both PCCE and standard colonoscopy. | within 7 days
Grading of the bubbles interference at the colon for PCCE. | Within 7 days
Percentage of excreted colon capsules | Within 7 Days
PCCE transit time from ingestion to excretion and colon transit time | Within 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Josef Sung, Prof., Principal Investigator — Chinese University of Hong Kong
Locations (3):
- Chinese university of Hong Kong, Princes of Walses Hospital, Hong Kong, Hong Kong
- Department of Medicine, National University Hospital, Singapore, Singapore
- Department of Internal Medicine & Health Management Center, National Taiwan University Hospital, Taipei, Taiwan